CLINICAL TRIAL: NCT02379390
Title: Phase II, Randomized, Open-label, Multicenter Study in Chemotherapy-naïve Metastatic Castration-Resistant Prostate Cancer (mCRPC) Patients Who Have PRIMary Resistance to Abiraterone Acetate or Enzalutamide Treatment Comparing the Anti-tumor Effect of CABazitaxel to Alternative Androgen Receptors (AR) Targeted Therapy
Brief Title: Cabazitaxel Versus the Switch to Alternative AR Targeted Therapy Enzalutamide or Abiraterone in Metastatic Castration-Resistant Prostate Cancer (mCRPC) Primary Resistant Patients to Abiraterone or Enzalutamide
Acronym: PRIMCAB
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unsatisfactory patient accrual
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS14022; U1111-1160-6008 (Other: UTN)
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — cabazitaxel; enzalutamide; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cabazitaxel (Experimental): Participants received Cabazitaxel 25 mg/m^2, intravenously for 1 hour along with prednisone 10 mg orally on Day 1 of every treatment cycle (each cycle was of 3 weeks) until disease progression, unacceptable toxicity, or participant's refusal of further study treatment.
  Interventions: Drug: Cabazitaxel XRP6258; Drug: Prednisone
- Abiraterone acetate or Enzalutamide (Active Comparator): Participants received abiraterone acetate 1000 mg (4 tablets of 250 mg), orally once daily along with prednisone 5 mg, orally twice daily from Day 1 to 21 in each treatment cycle (each cycle was of 3 weeks) or enzalutamide 160 mg, orally, until disease progression, unacceptable toxicity, or participant's refusal of further study treatment.
  Interventions: Drug: Ezalutamide; Drug: Abiraterone acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Cabazitaxel XRP6258
  Other Names: Jevtana
  Arms: Cabazitaxel
Drug: Ezalutamide
  Other Names: Xtandi
  Arms: Abiraterone acetate or Enzalutamide
Drug: Abiraterone acetate
  Other Names: Zytiga
  Arms: Abiraterone acetate or Enzalutamide
Drug: Prednisone

SUMMARY:
Primary Objective:

To demonstrate the superiority in term of radiographic Progression-Free Survival (rPFS) of cabazitaxel at at 25 milligram per meter square (mg/m^2) plus prednisone (Arm A) versus either enzalutamide at 160 milligram (mg) once daily or abiraterone acetate at 1000 mg once daily plus prednisone (Arm B) in chemotherapy-naïve participants with metastatic Castration-Resistant Prostate Cancer (mCRPC) who have disease progression while receiving androgen receptor (AR) targeted therapy (abiraterone plus prednisone or enzalutamide) within 12 months of treatment initiation (≤12 months).

Secondary Objective:

* To compare efficacy for:
* Prostate-specific antigen (PSA) response rate and Time to PSA progression (TTPP).
* Progression Free Survival (PFS).
* Overall Survival (OS).
* Tumor response rate in participants with measurable disease (RECIST 1.1)
* Pain response and time to pain progression.
* Symptomatic skeletal events (SSE) rate and time to occurrence of any SSE.
* To analyze messenger ribonucleic acids (mRNAs) including androgen-receptor splice variant 7 messenger RNA (AR-V7) as a biomarker in Circulating Tumor Cells (CTCs).
* To evaluate safety in the 2 treatment arms.

DETAILED DESCRIPTION:
The duration of the study per participant was approximately 2 years. Each participant was treated until radiographic disease progression, unacceptable toxicity, or participants refusal of further study treatment, and each participant was followed after completion of study treatment until death, study cutoff date, or withdrawal of participant consent.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of histologically or cytologically confirmed prostate adenocarcinoma.
* Metastatic disease.
* Progressive disease (PD) while receiving AR targeted therapy with abiraterone acetate or enzalutamide within 12 months of treatment initiation (≤12 months) by at least one of the following:
* Progression in measurable disease Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Appearance of 2 or more new bone lesions according to Prostate Cancer Working Group 2 (PCWG2).
* Rising PSA defined (PCWG2) as at least two consecutive rises in PSA to be documented over a reference value (measure 1) taken at least one week apart.
* A PSA value of at least 2 nanogram/milliliter (ng/mL) is required at study entry.
* Effective castration (serum testosterone levels ≤0.5 ng/mL).
* Prior AR targeted therapy (abiraterone acetate or enzalutamide) must be stopped at least 2 weeks before study treatment.
* Signed written informed consent.

Exclusion criteria:

* Prior chemotherapy for prostate cancer, except estramustine and except adjuvant/neoadjuvant treatment completed >3 years ago. No further anti-cancer therapy after the previous AR targeted therapy and before inclusion. Prior docetaxel in hormone sensitive setting is allowed if completed >1 year before randomization. Prior immunotherapy is allowed.
* Less than 28 days elapsed from prior treatment with immunotherapy, radiotherapy, or surgery to the time of randomization.
* Adverse events (excluding alopecia and those listed in the specific exclusion criteria) from any prior anticancer therapy of grade >1(National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v4.0) at the time of randomization.
* Eastern Cooperative Oncology Group (ECOG) performance status >1.
* History of brain metastases, uncontrolled spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease.
* Prior malignancy. Adequately treated basal cell or squamous cell skin or superficial (pTis, pTa, and pT1) bladder cancer are allowed, as well as any other cancer for which treatment has been completed ≥5 years ago and from which the patient has been disease-free for ≥5 years.
* Participation in another clinical trial and any concurrent treatment with any investigational drug within 30 days prior to randomization.
* Acquired immunodeficiency syndrome (AIDS)-related illnesses or known Human immunodeficiency virus (HIV) disease requiring antiretroviral treatment.
* Any severe acute or chronic medical condition including uncontrolled diabetes mellitus, severe renal impairment, history of cardiovascular disease (uncontrolled hypertension, arterial thrombotic events in the past 6 months, congestive heart failure, severe or unstable angina pectoris, recent myocardial infraction within last 6 months or uncontrolled cardiac arrhythmia), which could impair the ability of the patient to participate to the study or interfere with interpretation of study results, or patient unable to comply with the study procedures.
* Participants with reproductive potential who do not agree to use accepted and effective method of contraception during the study treatment period and up to 6 months after the last administered dose. The definition of "effective method of contraception" will be based on the Investigator's judgment.
* Known allergies, hypersensitivity or intolerance to prednisone or excipients of abiraterone acetate or enzalutamide. History of hypersensitivity to docetaxel or polysorbate 80.
* Known history of mineralocorticoid excess or deficiency (not applicable to participants who have already been treated with abiraterone acetate in first line before inclusion).
* History of seizure, underlying brain injury with loss of consciousness, transient ischemic attack within the past 12 months, cerebral vascular accident, brain arteriovenous malformation or the use of concomitant medications that may lower the seizure threshold (not applicable to participants who have already been treated with enzalutamide in first line before inclusion).
* Unable to swallow a whole tablet or capsule.
* Inadequate organ and bone marrow function as evidenced by:
* Hemoglobin <10.0 g/dL.
* Absolute neutrophil count <1.5 x 10^9/L.
* Platelet count <100 x 10^9/L.
* Aspartate aminotransferase (AST) and/or Alanine aminotransferase (ALT) >1.5 x Upper limit of normal (ULN).
* Total bilirubin >1.0 x ULN.
* Potassium <3.5 mmol/L.
* Serum albumin <3.0 g/dL.
* Child-Pugh Class B and C.
* Contraindications to the use of corticosteroid treatment.
* Symptomatic peripheral neuropathy grade ≥2 NCI CTCAE v4.0.
* Concomitant vaccination with yellow fever vaccine.

The above information was not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-06-17 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (24):
- United States (14):
  - Investigational Site Number 840030, Muscle Shoals, Alabama
  - Investigational Site Number 840024, Anchorage, Alaska
  - Investigational Site Number 840028, Anaheim, California
  - Investigational Site Number 840004, Sacramento, California
  - Investigational Site Number 840002, Boca Raton, Florida
  - Investigational Site Number 840027, Lakeland, Florida
  - Investigational Site Number 840006, Port Saint Lucie, Florida
  - Investigational Site Number 840015, Ottawa, Illinois
  - Investigational Site Number 840001, Covington, Louisiana
  - Investigational Site Number 840017, Metairie, Louisiana
  - Investigational Site Number 840012, Rockville, Maryland
  - Investigational Site Number 840026, Omaha, Nebraska
  - Investigational Site Number 840022, Canton, Ohio
  - Investigational Site Number 840016, Myrtle Beach, South Carolina
- Canada (10):
  - Investigational Site Number 124003, Edmonton
  - Investigational Site Number 124010, Greenfield Park
  - Investigational Site Number 124005, Hamilton
  - Investigational Site Number 124004, London
  - Investigational Site Number 124002, Montreal
  - Investigational Site Number 124006, Montreal
  - Investigational Site Number 124007, Ottawa
  - Investigational Site Number 124009, Québec
  - Investigational Site Number 124008, Saskatoon
  - Investigational Site Number 124001, Vancouver

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted at 6 active centers in United States and Canada. A total of 8 participants were enrolled between 17 June 2015 to 13 Mar 2016. Total 15 participants were screened, out of which 7 were screen failures and 8 were randomized and treated in the study. Study was terminated early due to very low recruitment rate in both countries involved.
Pre-assignment Details: Participants were randomized to receive either chemotherapy (cabazitaxel) or antiandrogen receptor targeted therapy (abiraterone or enzalutamide were assigned based on previous Androgen receptor [AR] targeted treatment in which participants previously treated with abiraterone were treated with enzalutamide and vice versa due to resistance).
Groups:
- Cabazitaxel: Participants received Cabazitaxel 25 milligrams per meter square (mg/m^2), intravenously for 1 hour on Day 1 of each cycle (each cycle was of 3 weeks), plus prednisone 10 milligrams (mg) orally given daily until radiographic disease progression, unacceptable toxicity, or participant's refusal of further study treatment.
- Abiraterone Acetate or Enzalutamide: Participants received abiraterone acetate 1000 mg (4 tablets of 250 mg), orally continuously once daily along with prednisone 5 mg, orally twice daily from Day 1 to 21 in each treatment cycle (each cycle was of 3 weeks) or enzalutamide 160 mg, orally continuously once daily from Day 1 to Day 21 in each treatment cycle (each cycle was of 3 weeks), until radiographic disease progression, unacceptable toxicity, or participant's refusal of further study treatment.
Period: Overall Study
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Started | 4 | 4
Completed (Participant with Disease Progression were counted as completed.) | 2 | 2
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Investigator's decision | 1 | 0
Not completed — Study Termination | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who were exposed to at least one dose of study treatment.
Groups:
- Cabazitaxel: Participants received Cabazitaxel 25 mg/m^2, intravenously for 1 hour on Day 1 of each cycle (each cycle was of 3 weeks), plus prednisone 10 mg orally given daily until radiographic disease progression, unacceptable toxicity, or participant's refusal of further study treatment.
- Total: Total of all reporting groups
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression-Free Survival (rPFS)
Description: rPFS was defined as the time from randomization to the first occurrence of radiological tumor progression using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or progression of bone lesions using prostate cancer working group 2 (PCWG2) criteria or death due to any cause.
Time Frame: Baseline until tumor progression or bone lesion progression or death due to any cause (maximum duration: 1059 days)
Population: Planned analysis could not be performed due to early study termination.
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Prostate Specific Antigen (PSA) Response
Description: PSA response was defined as decline of serum PSA from baseline by >= 50 percent (%).
Time Frame: Baseline up to PSA progression or death due to any cause (maximum duration: 1059 days)
Population: Planned analysis could not be performed due to early study termination.
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS: time interval between date of randomization to first documentation of tumor progression as per RECIST 1.1.
Time Frame: Baseline upto progression or death due to any cause (maximum duration: 1059 days)
Population: Planned analysis could not be performed due to early study termination.
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Survival
Description: Overall Survival was defined as the time interval from the date of randomization to the date of death due to any cause.
Time Frame: Baseline until death or study cut-off date, whichever was earlier (maximum duration: 1059 days)
Population: Planned analysis could not be performed due to early study termination.
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to PSA Progression
Description: Time to PSA progression was defined as the time interval between the date of randomization and the date of first documented PSA progression as per PCWG2 criteria.
Time Frame: Baseline up to PSA progression or death due to any cause (maximum duration: 1059 days)
Population: Planned analysis could not be performed due to early study termination.
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants Achieving Tumor Response
Description: Tumor response was defined as either a partial response (PR) or complete response (CR) according to the RECIST 1.1.
Time Frame: Baseline up to disease progression or death due to any cause (maximum duration: 1059 days)
Population: Planned analysis could not be performed due to early study termination.
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Duration of Tumor Response
Description: Duration of tumor response was defined as the time between the first evaluation at which the tumor response criteria were met and the first documentation of tumor progression.
Time Frame: Baseline up to disease progression or death due to any cause (maximum duration: 1059 days)
Population: Planned analysis could not be performed due to early study termination.
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Pain Response Using Brief Pain Inventory-Short Form (BPI-SF) for Pain Intensity Score
Description: Pain response was analyzed using the brief pain inventory-short form (BPI-SF).
Time Frame: Baseline until the end of study (maximum duration: 1059 days)
Population: Planned analysis could not be performed due to early study termination.
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time to Pain Progression
Description: Time to pain progression was defined as the time interval between the date of randomization and the date of the first documented pain progression.
Time Frame: Baseline until disease progression, start of another anticancer therapy or study cut off, whichever came first (maximum duration: 1059 days)
Population: Planned analysis could not be performed due to early study termination.
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percentage of Participants With Symptomatic Skeletal Event (SSE)
Description: SSE was the occurrence of a new symptomatic pathological fracture, or the use of external beam radiation to relieve bone pain, or the occurrence of spinal cord compression, or tumor-related orthopedic surgical intervention.
Time Frame: Baseline until the end of study (maximum duration: 1059 days)
Population: Planned analysis could not be performed due to early study termination.
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Time to Occurrence of Any Symptomatic Skeletal Events (SSE)
Description: Time to SSE was defined as the time interval between the date of randomization and the date of the occurrence of the first event defining a SSE, whichever is earlier.
Time Frame: Baseline up to occurrence of the first event defining a SSE (maximum duration: 1059 days)
Population: Planned analysis could not be performed due to early study termination.
Arm/Group | Cabazitaxel | Abiraterone Acetate or Enzalutamide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline until the end of study (maximum duration: 1059 days)
Groups:
- Enzalutamide or Abiraterone: Participants received abiraterone acetate 1000 mg (4 tablets of 250 mg), orally continuously once daily along with prednisone 5 mg, orally twice daily from Day 1 to 21 in each treatment cycle (each cycle was of 3 weeks) or enzalutamide 160 mg, orally continuously once daily from Day 1 to Day 21 in each treatment cycle (each cycle was of 3 weeks), until radiographic disease progression, unacceptable toxicity, or participant's refusal of further study treatment.
- Abiraterone: Participants received abiraterone acetate 1000 mg (4 tablets of 250 mg), orally continuously once daily along with prednisone 5 mg, orally twice daily from Day 1 to 21 in each treatment cycle (each cycle was of 3 weeks) until radiographic disease progression, unacceptable toxicity, or participant's refusal of further study treatment.
- Enzalutamide: Participants received enzalutamide 160 mg, orally continuously once daily from Day 1 to Day 21 in each treatment cycle (each cycle was of 3 weeks), until radiographic disease progression, unacceptable toxicity, or participant's refusal of further study treatment.
Arm/Group | Cabazitaxel | Enzalutamide or Abiraterone | Abiraterone | Enzalutamide
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/4 | 0/1 | 2/3
Other Adverse Events (participants affected / at risk) | 3/4 | 2/4 | 1/1 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabazitaxel (N=4) | Enzalutamide or Abiraterone (N=4) | Abiraterone (N=1) | Enzalutamide (N=3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabazitaxel (N=4) | Enzalutamide or Abiraterone (N=4) | Abiraterone (N=1) | Enzalutamide (N=3)
Increased Tendency To Bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood Swings (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT02379390/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT02379390/SAP_001.pdf